CLINICAL TRIAL: NCT04378283
Title: Prospective Evaluation of Topical Anesthesia in Children
Acronym: LET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Michael Boettcher, PD Dr. Michael Boettcher, Universitätsklinikum Hamburg-Eppendorf
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHHamburgEppendorf_LET
Record Dates: First submitted 2016-05-16; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Skin Lacerations
MeSH Terms: interventions — Lidocaine; Epinephrine; Lidocaine, Prilocaine Drug Combination; Anesthetics; Wound Healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LET as topical anesthetic for wound repair. (Experimental): LET gel (lidocaine 4%, epinephrine 0.1%, and tetracaine 0.5%) is a topical anesthetic that is routinely used before laceration repair.
  Interventions: Drug: LET gel (lidocaine 4%, epinephrine 0.1%, and tetracaine 0.5%)
- EMLA plus infiltration as anesthetic for wound repair. (Active Comparator): EMLA ("eutectic mixture of local anesthetics") with subsequent lidocaine infiltration. EMLA is a mixture of lidocaine (2.5%) and prilocaine (2.5%) in a cream base.
  Interventions: Drug: EMLA plus infiltration as anesthetic for wound repair.

INTERVENTIONS:
Drug: LET gel (lidocaine 4%, epinephrine 0.1%, and tetracaine 0.5%) — The study is designed to evaluate topical anesthetics
  Arms: LET as topical anesthetic for wound repair.
Drug: EMLA plus infiltration as anesthetic for wound repair. — EMLA plus infiltration as anesthetic for wound repair.
  Arms: EMLA plus infiltration as anesthetic for wound repair.

SUMMARY:
This study is designed to assess efficacy and comfort of LET solution vs. EMLA cream and topical infiltration of lidocaine.

DETAILED DESCRIPTION:
Pain caused by repair of torn skin is usually an unpleasant experience for pediatric patients. Analgesia or pain control is conventionally achieved by local anaesthetic infiltration. Local anaesthetics are a class of drugs that interrupt the transmission of electrical impulses along sensory nerves by inactivating sodium channels (Eidelman et al., 2011). However, the infiltration of local anaesthetics, which involves injecting the medication into the skin, may itself cause significant pain and fear in children (Kundu and Achar, 2002, Boettcher et al., 2012).

Pain management has been increasingly recognized as an element of high quality patient care, yet studies have shown deficiencies in pediatric emergency department (PED) pain management in children (Lawton and Hadj, 2014, Fein et al., 2012). Resolution of pain and perception of pain have been documented as one of the top indicators of patient and parent satisfaction and measure of quality of care in the PED (Magaret et al., 2002). Children are particularly susceptible to pain, even when caused by simple procedures (Boettcher et al., 2012). Well-managed pain has been associated with faster recoveries, fewer complications, and decreased use of health care resources (Zhu et al., 2012).

LET gel (lidocaine 4%, epinephrine 0.1%, and tetracaine 0.5%) is a topical anesthetic that is routinely used before laceration repair. LET gel offers many advantages for repair of tissue laceration including epinephrine-induced vasoconstriction, promotion of dry surfaces required for tissue adhesive laceration repair, and reduction of discomfort (MacLean et al., 2007). Topical anesthetics have been shown to improve procedural success rates and reduce procedural times, likely due to decreased patient movement and pain reduction (Taddio et al., 2005). LET has been shown to significantly reduce the need for injecting local anesthetics to the wound site, which is a cause of much anxiety and pain in children (Taddio et al., 2005, Singer and Stark, 2001).

In many PED - as in our department - LET solution and EMLA pretreatment and subsequent lidocaine infiltration are used depending on the personal experience and preference of the physician. The objective of this study is to determine if LET solution is as effective as EMLA and lidocaine infiltration in terms of comfort and effectiveness.

Primary Hypothesis:

LET solution is as effective as EMLA and lidocaine infiltration in controlling pain.

Secondary Hypothesis:

LET solution is superior to EMLA and lidocaine infiltration in terms of comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Chronological age above 3 and below 18 years
2. Dermal laceration that needs surgical repair
3. Signed informed consent by the parent or guardian of the patient

Exclusion Criteria:

* Skin laceration of nose tip, fingers, genitalia

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Pain during skin repair | 2 weeks
  Pediatric pain scale

SECONDARY OUTCOMES:
Infections during skin repair | 2 weeks
  Purulent discharge from the surgical site Purulent discharge from wound or drain placed in wound Organisms isolated from aseptically obtained wound culture Must be at least one of the signs and symptoms of infection - pain or tenderness, localised swelling, or redness/heat.
Speed during skin repair | 2 weeks
  Time from start until wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boettcher, MD PhD, Principal Investigator — UKE Medical School
Locations (1):
- UKE Medical School, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No